CLINICAL TRIAL: NCT06636292
Title: Using Virtual Reality Distraction and Disassociation (VRDD) in Adult Gastrointestinal Endoscopy
Brief Title: VRDD in Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Collaborators: EvoEndo, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 323884
Record Dates: First submitted 2024-08-23; First posted 2024-10-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Patient Satisfaction; Patient Acceptance of Health Care
Keywords: virtual reality; upper gastrointestinal endoscopy; transnasal endoscopy
MeSH Terms: conditions — Patient Satisfaction; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients having sedated TNE or any oesophagogastroduodenoscopy (OGD) (Active Comparator): Patients who are only recruited to Stage 1 of study to experience VRDD pre-endoscopy.
  Interventions: Device: Virtual Reality Distraction and Disassociation (VRDD) Stage 1
- Patients having unsedated TNE (Active Comparator): Patients who are recruited to both Stages 1 and 2 of study to experience VRDD pre-endoscopy and during endoscopy.
  Interventions: Device: Virtual Reality Distraction and Disassociation (VRDD) Stage 1&2

INTERVENTIONS:
Device: Virtual Reality Distraction and Disassociation (VRDD) Stage 1 — Participants wear a VR headset which plays VR content/material pre- endoscopy only.
  Arms: Patients having sedated TNE or any oesophagogastroduodenoscopy (OGD)
Device: Virtual Reality Distraction and Disassociation (VRDD) Stage 1&2 — Participants wear a VR headset which plays VR content/material pre- endoscopy and during endoscopy.
  Arms: Patients having unsedated TNE

SUMMARY:
The demand for gastrointestinal (GI) endoscopy is rising year by year and improving the patient's experience of having the procedure has become an important aim. A lot of work has been done in recent years on how to improve a patient's experience during GI endoscopy such as improving endoscopy and communication skills. Due to the increasing popularity of Virtual Reality (VR) in the gaming world, VR equipment have been used in children as a safe and effective distraction method during GI endoscopy, removing the need for them to have general anaesthesia for their procedure. This has been thought of as an option for the adult patients which would also save them from requiring sedation for their endoscopy procedure.

This is a pilot feasibility study (small scale preliminary study) carried out at a single hospital site with a dedicated GI endoscopy service. We intend to find out whether the VR headset that is used is tolerated and accepted by adult patients during their endoscopy procedure. This has been shown to be a cheaper option compared to giving sedation drugs or general anaesthesia as well. If adult patients can accept this option, we are hoping to investigate in future larger studies whether they could potentially use this as a distraction method to help improve their experience of undergoing GI endoscopy. Any adult patient who is having an upper GI endoscopy could be potentially eligible. Their endoscopy procedure forms part of their clinical care whereas the research component involves them wearing the VR headset before and/or during their procedure. Their experience of undergoing upper GI endoscopy and wearing the VR headset will be measured using a series of questionnaires.

DETAILED DESCRIPTION:
Study design:

This is a small scale preliminary study (pilot feasibility study) which is split into 2 stages. In the first stage, it will investigate if the VRDD equipment is acceptable for an adult patient to use prior to any upper GI endoscopy, including sedated and unsedated procedures. In the second stage, it will investigate whether the VRDD equipment is acceptable specifically for adult patients who have unsedated transnasal endoscopy (TNE). This study will be carried out by the research team who are based at one National Health Service (NHS) hospital i.e. South Tyneside District Hospital in the United Kingdom. The study is funded by EvoEndo, Inc which is based in Colorado, USA (provision of VR equipment). The investigators aim to recruit approximately 30 participants to the study, all of whom will have been referred for an upper GI endoscopy procedure for any clinical reason.

Once a patient has expressed their interest, they will be provided with a participant information sheet to read through. A research team member will be available to answer any queries. Patients who are keen to participate in the study will be asked to sign a consent form for them to be officially recruited into the study. This can be done a few days prior or on the day of their endoscopy procedure. It will be made clear to them that their endoscopy procedure will go ahead regardless of their participation in research because the procedure itself is part of standard clinical care and not research. They will need to sign a separate NHS consent form specifically for the upper GI endoscopy procedure which will be handled by the endoscopy team.

The VR equipment comprises of a headset which the participants will wear right before their procedure. It can play virtual reality images or videos from a mobile phone attached to the front of the headset. The VR content has been provided by the funding body (EvoEndo, Inc) which includes classic television programmes, sports programmes, movies, documentaries and children's entertainment.

Stage 1:

In Stage 1, participants will put on the VR headset before their endoscopy for approximately 10 minutes under supervision of a research team member. Once time is up, the VR headset will be removed and Stage 1 is complete. Participants will be provided with a few questionnaires that are relevant to this stage to complete in their own time.

They will be monitored for approximately another 10 minutes for any adverse effects before they proceed to their endoscopy procedure.

Stage 2:

This only involves patients who are having unsedated transnasal endoscopy. Patients who are having a gastroscopy will not progress to this stage.

For patients who choose to have transnasal endoscopy without sedation, the research team member will ask if they would like to proceed to Stage 2 of the study. This involves wearing the VR headset during their endoscopy. If they agree, it will be reattached onto them after all routine safety checks have been completed pre-endoscopy. The VR headset will remain on them for the duration of their endoscopy, unless they withdraw consent for using VRDD. After the endoscopy is completed, the VR headset will be removed for the participant to take home with them. They will be asked to remain in the endoscopy unit for approximately 10 minutes to allow any VRDD side effects to resolve before they leave. However, if they choose to not proceed onto Stage 2, this indicates the end of their participation in the study. The endoscopy procedure will still go ahead because it is part of standard clinical care.

Patients who have sedation for endoscopy will not be eligible to participate in Stage 2 of the study.

Participants can withdraw consent at any point. If they decide to withdraw study participation before the endoscopy, they would be asked to contact the research team about it. If they decide to withdraw study participation during their endoscopy, they would be advised to inform the endoscopy nurses who will inform the research team. A research team member will then remove the VR headset. Endoscopy will continue in both these scenarios because it is part of standard care. If participants withdraw consent for endoscopy at any point, they automatically become ineligible for the study.

Participants will not be able to remove their VR headset without assistance. If they confirm that they want to remove their headset, they can notify the endoscopy nurses who will ask a research team member who is outside the endoscopy room to come in to remove it. This would be considered a withdrawal of consent for ongoing study participation.

Data collection:

All participants from both stages will be asked to complete the VRDD questionnaire which assesses their experience of using the VR headset. In addition, they will be asked to complete the Newcastle ENDOPREM™ (assess patient experience of having upper GI endoscopy) and the modified Group Health Association of America-9 (mGHAA-9) survey. Participants can complete the questionnaires either on the day after they have had their endoscopy or at home. Completed questionnaires can be posted back to the research department in pre-paid envelopes which are marked confidential. All participants are strongly encouraged to do this within 3-4 days of their endoscopy and the latest within 7 days to allow an accurate recollection and reflection of their experiences. They may be contacted via telephone by a research team member on day 4, day 8 and day 10 after the endoscopy as a reminder if it is necessary to do so. The research team will be responsible for ensuring that all questionnaires have been received from the participants.

The end of study is defined as the date of the last visit of the last participant and by completion of data collection from the questionnaires.

It is anticipated that the investigators will need approximately 2-3 months to meet the recruitment target. Data collected from the questionnaire responses will be analysed and summarised by the research team. No follow-up research appointments are required from the study participants.

ELIGIBILITY:
Inclusion criteria:

• Referred with a clinical need for upper GI endoscopy (either transnasal or per oral route) on an elective basis.

Exclusion criteria:

* Planned therapeutic procedures (including but not limited to polypectomy, balloon dilatation, stenting).
* Uncorrected visual or auditory impairments or adaptions (e.g. spectacles) that make wearing the VR equipment difficult.
* Cognitive impairment or learning disabilities.
* Epilepsy.
* Balance disorders.
* Referred for urgent or emergency GI endoscopy.

Withdrawal criteria:

* Patients who withdraw consent from study participation.
* Patients who withdraw consent for having the endoscopy procedure.
* Patients who request to remove the VRDD equipment during Stages 1 or 2 of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Acceptability and tolerability of VRDD in adult patients using VRDD questionnaire | 2-3 months
  The acceptability and tolerability of using VRDD in all adult patients referred for upper GI endoscopy, measured on Likert scale via VRDD questionnaire

SECONDARY OUTCOMES:
Acceptability of VRDD in unsedated TNE using VRDD questionnaire | 2-3 months
  The acceptability of using VRDD in adult patients who undergo unsedated TNE, measured on Likert scale via VRDD questionnaire
Patient experience of using VRDD while having unsedated TNE using Newcastle ENDOPREM™ and mGHAA-9 questionnaires | 2-3 months
  The patient experience of undergoing unsedated TNE while using VRDD, measured on Likert scale via Newcastle ENDOPREM™ and mGHAA-9 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Phey Shen Lee, Study Chair — South Tyneside and Sunderland NHS Foundation Trust
Locations (1):
- South Tyneside District Hospital, South Shields, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No